CLINICAL TRIAL: NCT02471690
Title: A Randomized, Double-Blind, Single Center Cohort Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a New Formulation of a Single 1200MG IV Dose of Oritavancin in Healthy Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a New Formulation of Oritavancin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MDCO-ORI-15-01
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — oritavancin; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oritavancin (Active Comparator): IV -Single Dose - 1200 mg Oritavancin
  Interventions: Drug: Oritavancin
- Placebo (Placebo Comparator): 250 mL Dextrose 5% in Water
  Interventions: Drug: Dextrose

INTERVENTIONS:
Drug: Oritavancin — IV - Single dose 1200 mg Oritavancin
  Other Names: Orbactiv
  Arms: Oritavancin
Drug: Dextrose — D5W 5% in Water
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The protocol describes a double-blind study to evaluate the Pharmacokinetics and safety of a new formulation of oritavancin by adjusting infusion time, concentration and reconstitution/administration solutions, of a single 1200 mg intravenous (IV) infusion of oritavancin

DETAILED DESCRIPTION:
Oritavancin has been approved in the United States for the treatment of adult patients with acute bacterial skin and skin structure infections (ABSSSIs) caused or suspected to be caused by susceptible isolates of designated Gram-positive microorganisms. This is a Phase I, single center, double-blind, study evaluating the PK and safety of a new formulation of oritavancin by adjusting infusion time, concentration and reconstitution/administration solutions, of a single 1200 mg intravenous (IV) infusion of oritavancin in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent before initiation of any study related procedures.
2. Healthy male or female between the ages of 18 and 65 years, inclusive.
3. Body mass index (BMI) < 45 kg/m^2.
4. Subject is in good health based on medical history and physical examination findings and has no clinically meaningful safety laboratory abnormalities (CBC, blood chemistry, and urinalysis) or 12 lead ECG results, as assessed by the PI.
5. Vital signs (BP, pulse and temperature) measured at screening/baseline must be within the following ranges: SBP ≥90 to ≤150 mm Hg, DBP ≥45 to ≤90 mm Hg; Heart Rate ≥ 40 to ≤90 bpm (taken after resting in a supine position for at least 5 minutes).
6. Willing to avoid all medications (other than the study drug and acetaminophen/paracetamol for minor aches/pains) during the study. This includes prescription and non-prescription medications, vitamins, herbal supplements, and nutraceuticals.
7. Non-smoker and is willing to abstain from alcohol/illegal drug use for the duration of the study.
8. If the female subject is surgically sterile, postmenopausal, or, if of childbearing potential, agrees to use at least 2 highly-effective methods of birth control (e.g. prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods, abstinence) or male partner sterilization alone for the duration of the study until 60 days after study drug administration.

Exclusion Criteria:

1. Has any condition, including findings in the medical history or in pre-study assessments that constitutes a risk or a contraindication for the participation in the study or completing the study.
2. Female subjects of childbearing potential that have a positive test result for human chorionic gonadotropin (hCG) at screening.
3. Female subjects who are nursing.
4. Positive urine test for alcohol and/or for drugs of abuse at screening.
5. Has a history or presence of alcohol/drug abuse within 2 years. Alcohol abuse is defined as regularly consuming >3 units/day (21 units per week for men), >2 units/day (14 units/week) for women. 1 unit of alcohol is defined as a can of 4% beer (330 mL), approximately 190 mL of 6-7% beer (malt liquor), a glass of 40% spirits (30 mL), or a glass of wine (100 mL).
6. History of hypersensitivity to drugs with a similar chemical structure (i.e. glycopeptide antibiotics) to oritavancin or any of its excipients.
7. Blood or plasma donation within the past 2 months.
8. Subjects who participated in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days or 5 half-lives, whichever is longer, prior to screening and/or unwilling to allow at least two months before participation in another drug trial following the current trial.
9. Treatment with any prescription or OTC drugs, within 2 weeks or 5 half-lives, whichever is longer, or herbal nutritional supplements within 2 weeks of screening, with the exception of acetaminophen/paracetamol for minor aches/pains. Subjects will not be allowed to receive medications for the duration of the study (except the above mentioned acetaminophen/paracetamol). Birth control or other hormone replacement is also permitted as long as it has been taken at a stable dose for at least three months before the screening visit and remains stable for the duration of the study.
10. Males who are unwilling to practice abstinence or use an acceptable method of birth control during the entire study period (i.e. condom with spermicide).
11. Subjects that have any surgical or medical condition that could interfere with the administration of the study drug.
12. Subjects that have known active hepatitis B or C, or human immunodeficiency virus (HIV) infection or has known immune deficiency disease at screening.
13. Subjects that have any condition that would confound or interfere with the assessment of safety.
14. Subjects that have poor IV access as determined by the investigator.
15. Prior exposure to Oritavancin alone or in combination with another product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability: AEs/SAEs | From Consent up to 14 days following termination of the study drug infusion.
  A composite measure of the number and types of AE/SAEs encountered and relationship to time of dosing
Safety & Tolerability: clinical safety laboratory results | From Consent up to 14 days following termination of the study drug infusion.
  A composite measure of multiple laboratory results assessing the clinical significance of any changes from baseline
Safety & Tolerability: vital sign measurements | From Consent up to 14 days following termination of the study drug infusion.
  A composite of multiple vital sign measurements, assessing the clinical significance of any changes from baseline
Safety & Tolerability: ECGs | From Consent up to 14 days following termination of the study drug infusion.
  A composite of multiple ECG measurements, assessing the clinical significance of any changes from baseline
Safety & Tolerability: physical examination findings | From Consent up to 14 days following termination of the study drug infusion.
  A composite of multiple physical examination findings, assessing the clinical significance of any changes from baseline

SECONDARY OUTCOMES:
PK parameters: Cmax and area under the plasma concentration-time curve | From pre-dose until 168 hours from last dose
  maximum measured plasma concentration
PK parameters: AUC | From pre-dose until 168 hours from last dose
  AUC from time zero to the time of the last measurable concentration
PK parameters: t1/2 | From pre-dose until 168 hours from last dose
  elimination half life
PK parameters: volume of distribution [Vz] and CL] | From pre-dose to 168 hours from last dose
  Volume of distribution
PK parameters: tmax | From pre-dose to 168 hours from last dose
  Time to Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States